CLINICAL TRIAL: NCT03576872
Title: The GI Binder: A Psychoeducational Intervention for Gastrointestinal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Theresa Jabaley, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-241
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Gastro Intestinal Cancer
Keywords: Gastro Intestinal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychoeducational intervention (Experimental): * Psychoeducational will be conducted prior to chemotherapy.
  * Teach session will occur prior and during administration of chemo
  * A small quiz will be conducted to asses understanding of the educational binder
  Interventions: Other: Psychoeducational

INTERVENTIONS:
Other: Psychoeducational — Providing a binder of educational materials with nurse-led instruction in preparing pancreatic and colorectal cancer patients for chemotherapy

SUMMARY:
This research study is evaluating the use of a binder of educational materials with nurse teaching to prepare patients for chemotherapy

DETAILED DESCRIPTION:
This research study is being done to investigate the feasibility of providing a binder of educational materials with nurse-led instruction in preparing pancreatic and colorectal cancer patients at Dana Farber for chemotherapy. The investigators want to evaluate whether the binder is helpful and usable for patients; and its effect on knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write, and converse in English.
* 18 years or older
* Scheduled for a new chemotherapy start (intravenous) to treat adenocarcinoma of the pancreas or colorectal cancer

Exclusion Criteria:

* Enrolled in a clinical trial for chemotherapy
* Major psychological diagnoses that would limit participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
80% or higher rate of completing at least 3 of 4 nurse-led encounters with participants | 8 weeks

SECONDARY OUTCOMES:
An average positive direction of change scores between participants' pre- and post- knowledge scores | 8 weeks
Average score of 24 or higher on the adapted Acceptability E-scale | 8 weeks
80% or higher on the index of rates for delivery of educational binders | 8 weeks
80% or higher on the index of rates for pre-chemotherapy teach sessions using the binders | 8 weeks
80% or higher on the index of rates for teach sessions using the binder on day 1 of chemotherapy | 8 weeks
80% or higher on the index of rates for follow-up phone calls and binder review prior to cycle 2 of chemotherapy | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Jabaley, PhD, RN, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No